PRINCIPAL INVESTIGATOR: A.P. Chen, MD, DCTD/NCI

STUDY TITLE: A Phase 2 Study of Cabozantinib (XL184), a Dual Inhibitor of MET and

VEGFR, in Patients with Metastatic Refractory Soft Tissue Sarcoma

**STUDY SITE:** NIH Clinical Center

Cohort: Standard

Consent Version: 03/18/2021

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

Alice P. Chen, Principal Investigator: 240-781-3320

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

# IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

# WHY IS THIS STUDY BEING DONE?

We are doing this study to try to develop better treatments for cancer. In this study, the experimental drug cabozantinib will be given to you. The purpose of this study is to find out if the drug is effective in a particular type of tumor called soft tissue sarcoma, which is what your doctor has diagnosed you with. We are trying to understand how these drugs work in soft tissue sarcomas. For that, this study will look at how cabozantinib may affect the levels of certain proteins in your tumor.

The use of cabozantinib in soft tissue sarcoma is experimental. **Cabozantinib** works by two mechanisms. Firstly, it acts by blocking the formation of new blood vessels in tumors, a process called angiogenesis. New blood vessels provide oxygen and nutrients to growing cancers, and blocking this process can cause cancer cells or the supporting blood vessels to stop growing. A

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 03/18/2021


drug that works by the same mechanism, pazopanib, has already been approved by the FDA for the treatment of patients with sarcoma. In laboratory studies, some drugs that block angiogenesis increase the production of c-MET in tumors, which helps cancer cells adapt to not having enough oxygen, so the tumor can keep growing. **Cabozantinib** also blocks c-MET in tumors. By both these mechanisms the ability of the sarcoma tumor cells to survive may be markedly reduced by the drug.

Although we hope this drug will decrease the size of your tumor, we cannot promise or predict the benefits of the treatment at this time. The drug used in this study has known side effects that will be reviewed with you by your medical team before you sign the consent form.

# WHY ARE YOU BEING ASKED TO TAKE PART IN THIS STUDY?

You are being asked to take part in this research study because you have advanced cancer that has progressed after receiving standard treatment, or for which no effective therapy exists.

# HAVE THESE DRUGS BEEN GIVEN TO OTHER PEOPLE?

**Cabozantinib** has been studied in many different cancer types like prostate cancer. So far, more than 1300 patients have received cabozantinib in clinical trials for different types of cancers.

# HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 55 patients will take part in this study at 4 centers across the United States.

#### DESCRIPTION OF RESEARCH STUDY

# WHAT WILL HAPPEN IF YOU TAKE PART IN THIS RESEARCH STUDY?

# Before you begin the study

You will need to have the following examinations, tests, or procedures to find out if you can be in the study. These tests are part of your regular cancer care and should be done by your health care team even if you do not join the study. If you have had them recently, they may not need to be repeated. This will be up to your study doctor.

If you decide that you would like to participate in this study, you will be asked to sign this consent form. You will then have the examinations, tests, and procedures listed below done to see if you can take part in the study (this is called the screening/baseline evaluation).

- Complete medical history.
- **Physical examination**, including height, weight, blood pressure, pulse, and temperature.
- **Standard blood tests** (requiring about 1 tablespoon of blood in total), which include measurement of your white blood cells, red blood cells, platelets, blood sugar and electrolytes, how your liver and kidneys work, and how well your blood clots.
- **Pregnancy test** in women who are able to become pregnant.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- **Urine tests:** A urine test will be done to check the level of protein excreted by your kidneys. Depending on the results of blood tests, you may be asked to collect your urine for 24 hours for further testing.
- **EKG** to check your heart.
- **CT scans** (a computerized x-ray examination) of your chest, abdomen, and pelvis to measure your tumor(s). Other imaging tests may be done as needed.
- **Pathology slides:** Before starting on the study, we will request tumor slides or blocks to confirm your diagnosis.

# **During the study**

If you are accepted and choose to take part, you will begin taking the study drug cabozantinib. Cabozantinib is taken by mouth. The study drug will be given in cycles. All cycles are 4 weeks (28 days) long.

Cabozantinib is taken 1 hour before or 2 hours after food. Each day that you take study drug, you will be asked to fill in a diary to show when you took the study drugs, how many pills you took, and report any side effects you may have had.

For some study procedures we will need you to come to the Clinical Center. You will also have tests performed because you are in the study to see how the study drug is affecting your body and to find out how your body handles the study drug. This will include imaging studies (for example, CT scans) to find out if your cancer has responded.

Clinical Center Visits: We will ask that you come to the Clinical Center for at least 2 days during the first cycle, and then at the beginning of each cycle after that (less often if you have been on study for more than one year). During the first cycle, you may be admitted to the Clinical Center for the first 2 days of drug administration to make it easier to perform study test and procedures to see how the drugs are affecting your body. If you develop any side effects, you may be asked to visit more often. Please see the study chart for more details.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# Standard procedures being done because you are in this study; these may be done more often because you are in the study:

- Clinic visit to ask how you are feeling and to evaluate you with a physical at the beginning of each cycle (up to 8 days before the start of each cycle; less often if you have been on study for more than one year).
- Vital signs and physical examination: will be performed during the clinic visits. We will ask that you buy a blood pressure monitor (the cost of may be reimbursed to you; discuss with your study team) and measure your own blood pressure at home at least once a day (preferably twice a day) throughout the study. You will record the readings in a diary. If your systolic blood pressure (top number) is ever more than 150 or your diastolic blood pressure (bottom number) more than 90, you should re-measure your blood pressure 1 to 4 hours later. If your systolic pressure is still greater than 150 or your diastolic blood pressure is still greater than 90, please contact your study team for instructions. You should also call the research team if you experience any symptoms of high blood pressure, such as chest pain, shortness of breath, headache, blood in the urine, or double vision.
- **Blood tests:** Measurement of your white blood cells, red blood cells and platelets, and measurements of your blood sugar, electrolytes, and how your liver and kidneys work will be done each time you are seen in the outpatient clinic. All of these blood tests combined will require 1-2 tablespoons (20-30 mL) of blood each time.
- Urine test to check urine protein will be done during the first cycle and then before you start each new cycle (less often if you have been on study for more than one year). You may need it more frequently if the study doctor thinks it is needed to check for signs of possible damage to your kidneys. Depending on the results of urine tests, you may be asked to collect your urine for 24 hours for further testing.
- CT scans or other imaging tests such as ultrasound (an examination using sound waves) or MRI (an examination using magnetic field and radio waves) that detect your tumor will be done every 2 cycles (about every 8 weeks; every 12 weeks if you have been on study for more than 1 year or every 16 weeks if on study for more than 3 years) while you are receiving treatment. This is done so that any benefit of the treatment can be determined, and so that if your cancer is not responding to the treatment, the study team can tell you and help you move to a different treatment program (discussed further below).

# Tests and procedures being done to see how the drug is affecting your body:

- Research blood samples: We will collect blood samples to help us find out if cabozantinib affects the levels of certain proteins. Blood will be collected before you first take the drug and on the first day of cycles 1 and 2 only. Please see the study chart for more details. The total blood for all these tests will be about 2 teaspoons.
- We will also be collecting optional blood samples to find out the effects of the drug on any tumor cells in your blood. Blood samples will be collected before you first take the drug, on the first day of cycle 1, and on the first day of every cycle for as long as you are on study (every 3 cycles if you have been on study for more than one year or every 4 cycles if more than 3 years). Each blood collection is about 2 teaspoons.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# STUDY CHART

The treatment is given over periods called cycles. All cycles are 4 weeks long. Treatment cycles will be repeated as long as you are tolerating the drugs and your cancer is either stable or getting better. Each cycle is numbered in consecutive order. The chart below shows what will happen during Cycle 1 and future cycles. The left-hand column shows the day in the cycle, and the right-hand column tells you what will happen on that day. This schedule shows what will happen to you after you sign the consent and start the study.

Cabozantinib should be taken with water at least 1 hour before or 2 hours after a meal. The drug tablets should be swallowed whole with water and may not be crushed or broken.

| Day | What to do and what will happen to you |
|---|---|
| Before starting study drugs | <ul> <li>Check in at Outpatient Clinic</li> <li>Get routine blood and urine tests</li> <li>Pregnancy test for women who are able to become pregnant</li> <li>Have a history taken of how you feel and undergo a physical examination including vital signs by a Health Care Provider (can be completed up to 8 days before the start of the study)</li> <li>CT or MRI scan will be done</li> <li>EKG will be done</li> <li>Research blood samples will be taken</li> </ul> |
| Cycle 1,<br>Day 1<br>Cycle 1,<br>Days 2 -28 | <ul> <li>Admitted to Clinical Center</li> <li>Begin taking cabozantinib 60 mg PO by mouth each day</li> <li>Research blood samples will be taken</li> <li>You will be asked to keep a record of pill consumption and any new symptoms</li> <li>Receive study diary</li> <li>Continue taking cabozantinib by mouth each day</li> </ul> |
| Cycles 2 and 3,<br>Day 1 | <ul> <li>Check in at Outpatient Clinic</li> <li>Return study diary</li> <li>Have a history taken of how you feel and undergo a physical examination including vital signs by a Health Care Provider (can be completed up to 8 days before the start of each new cycle)</li> <li>Pregnancy test for women who are able to become pregnant</li> <li>Get routine blood and urine tests (up to 8 days before)</li> <li>Get a routine EKG (up to 8 days before)</li> <li>Research blood samples will be taken</li> <li>Continue taking cabozantinib by mouth each day</li> </ul> |
| Cycles 2 and 3, | Continue taking cabozantinib by mouth each day |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| Day | What to do and what will happen to you |
|---|---|
| Days 2 -28 | |
| Cycle 4 onwards, D1 Clinic visits on D1 will be every 3 cycles (every 12 weeks) if you have been on study for more than one year or every 4 cycles (every 16 | <ul> <li>Continue taking cabozantinib by mouth each day</li> <li>Check in at Outpatient Clinic</li> <li>Return study diary</li> <li>Research blood samples will be taken on the first day of each cycle</li> <li>Have a history taken of how you feel and undergo a physical examination including vital signs by a Health Care Provider (can be completed up to 8 days before the start of each new cycle)</li> <li>Pregnancy test for women who are able to become pregnant</li> <li>Get routine blood and urine tests (up to 8 days before)</li> <li>EKG tests (up to 8 days before)</li> <li>CT scans to determine how your tumor is responding to the treatment</li> </ul> |
| weeks) if you have<br>been on study for<br>more than 3 years | will be done every 2 cycles (every 8 weeks; every 12 weeks if you have been on study for more than one year or every 16 weeks if more than 3 years) |

# RISKS OR DISCOMFORTS OF PARTICIPATION

# What side effects or risks can I expect from being in this study?

If you choose to take part in this study, there is a risk that the XL184 (cabozantinib) may not be as good as the usual approach for your cancer or condition at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The XL184 (cabozantinib) used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Here are important things to know about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it hard for you to have children.
- Some side effects may be mild. Other side effects may be very serious and even result in death

# PATIENT IDENTIFICATION Consent to Participate in a Clinical Research Study NIH-2977 (4-17) File in Section 4: Protocol Consent (1) Version Date: 03/18/2021  IRB NUMBER: 13C0044 

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

# **Drug risks**

The tables below show the most common and the most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you."

High blood pressure is one common side effect of cabozantinib. Your blood pressure will be closely watched while you are taking this drug. You will also be checking your blood pressure at home at least once a day (preferable twice a day) for the entire study. If you have high blood pressure while taking cabozantinib, your study doctor may recommend follow-up with your primary care physician and/or starting or increasing medication to lower your blood pressure.

Some patients on this study have experienced blood clots in the lungs, possibly related to the study drug. Let your doctor know immediately if you experience any shortness of breath or chest pain.

In addition, some patients on this study have experienced sepsis, or an infection in the bloodstream, possibly related to the study drug. This condition can cause fever, increased heart rate, increased breathing rate, and confusion. Sepsis can be life-threatening.

Grapefruit juice has been shown to affect how the body handles some drugs by blocking the activity of the body's cytochrome P450 (CYP450) system. CYP450 is important in breaking down substances in the body, including cabozantinib. Do not take grapefruit/grapefruit juice or Seville oranges while participating in this trial. Inform physician and study healthcare team about current medications including over the counter drugs, herbals, or natural medicines. We do not know if taking cabozantinib will cause other drugs you may be taking to work differently. It is very important that you talk to a member of the research team before beginning any new drugs, over-the-counter medications, vitamins, or alternative therapies.

Risks and side effects related to cabozantinib may include:

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving XL184 (cabozantinib), more than 20 and up to 100 may have:

- Diarrhea, nausea, vomiting
- Tiredness
- Weight loss, loss of appetite
- Changes in taste
- Redness, pain or peeling of palms and soles
- High blood pressure which may cause headaches, dizziness, blurred vision

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving XL184 (cabozantinib), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Pain
- Constipation, heartburn
- Dry mouth, skin
- Sores in the mouth which may cause difficulty swallowing
- Swelling of arms, legs
- Infection
- Bruising, bleeding
- Dehydration
- Muscle weakness
- Dizziness, headache
- Cough, shortness of breath
- Internal bleeding which may cause black tarry stool, blood in vomit, coughing up blood, or blood in urine
- Bleeding from multiple sites including the nose
- Changes in voice
- Hair loss, rash
- Change in hair color
- Blood clot which may cause swelling, pain, shortness of breath

#### RARE, AND SERIOUS

In 100 people receiving XL184 (cabozantinib), 3 or fewer may have:

- A tear or hole in internal organs that may require surgery
- Non-healing surgical site
- Damage to the jawbone which may cause loss of teeth
- Bleeding in the brain which may cause confusion
- Stroke which may cause paralysis, weakness
- Brain damage which may cause headache, seizure, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Lung collapse

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# Reproductive Risks

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how cabozantinib would affect your baby or your unborn child. If you are a woman who can become pregnant, or are the partner of a woman who can become pregnant, you will need to practice **two** effective forms of birth control before starting study treatment, during study treatment, and for 4 months after you finish study treatment. Your study team will talk with you about the kinds of birth control that can be used in this study.

If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [injections, or implants]: estrogen containing pills are not allowed due to the risk of blood clotting
- tubal ligation
- vasectomy

# **Side Effects of Blood Draw**

**Infrequent** (occurs in 1 to 10 out of 100 people): persistent pain and discomfort at the injection or needle insertion site as well as possible infection, bleeding, bruising, and soreness.

# What are the risks of radiation from being in the study?

# Potential Risks Related to Research-Related Imaging Studies:

During your participation in this research study, you may be exposed to radiation from up to 7 CT scans or FDG-PET/CT scans each year. The amount of radiation exposure from these procedures is equal to approximately 8 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT scans or FDG-PET/CT scans that you get in this study will expose you to roughly the same amount of radiation as 28 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.8 out of 100 (0.8%) and of getting a fatal cancer is 0.8 out of 100 (0.8%).

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# Potential Risks for FDG-PET/CT

In addition to the radiation risks described above, there is a chance of developing an allergic reaction from the FDG-PET contrast material, which may cause symptoms ranging from mild itching or a rash to severe difficulty breathing, shock or rarely, death. The contrast material may also cause kidney problems. The study doctors will do a blood test prior to the test to confirm that it is safe you to receive the contrast.

You may feel discomfort when the contrast material is injected. You may feel warm, flushed, get a metallic taste in your mouth or, rarely, may make you vomit or feel sick to your stomach.

The risks of IV insertion include temporary pain and bleeding or bruising at the site where the IV enters the skin. In placing the IV, there is a small chance of fluid leaking into the tissue surrounding the IV and infection, which may cause some swelling and discomfort. Rarely, the IV site may become infected, which might require treatment with antibiotics.

#### **Potential Risks for MRI**

People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

#### POTENTIAL BENEFITS OF PARTICIPATION

# Are there benefits to taking part in this study?

Taking part in this study may or may not make your health better. We do not know if you will receive personal, medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. You should discuss other treatment options with the study team and your home doctor before deciding to take part in this study. We do know that information from this study will help doctors learn more about these study drugs. This information will also help future cancer patients.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

# ALTERNATIVE APPROACHES OR TREATMENTS

# What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems, and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# RESEARCH SUBJECT'S RIGHTS

# What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in this study. If you decide to take part, you may leave the study at any time. No matter what decision you make, there will be no penalty to you, and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution if you are eligible and choose to participate in another trial. We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study. In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

# USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used.

Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

My specimens and data may be kept for use in research to learn about, prevent, or treat cancer or other health problems.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| Yes | No | Initials |
|-----|----|----------|

# COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

This study does not offer reimbursement for, or payment of, travel, lodging or meals.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays, or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs even if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.
- The study agent, cabozantinib, will be provided free of charge while you are participating in this study. Even though it is unlikely, there is a possibility that at some point the supply of study agents may run out, necessitating taking you off-study.
- Even though it is unlikely, the manufacturer may not continue to provide the cabozantinib to the NCI for some reason. If this would occur, other possible options are:
  - 1. You might be able to get cabozantinib from the manufacturer or your pharmacy but you or your insurance company may have to pay for it.
  - 2. If there is no cabozantinib available at all, no one will be able to get more and the study would close.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


• If a problem with getting cabozantinib occurs, your study doctor will talk to you about these options. Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.

# EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you
- if too many patients in the study experience severe side effects
- if you become pregnant

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to the Cancer Therapy Evaluation Program (CTEP) at the National Cancer Institute (NCI) or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

# **FOLLOW-UP**

You will be followed for 30 days after taking the last dose of study drug. We will call you after about 30 days to ask about any side effects that were ongoing when you stopped therapy, or any new side effects that might be related to the study therapy. If you have side effects that might be related to the study drugs that have not gotten better after 30 days, we will call you every 2 weeks until the side effects have become stable or gotten better. The follow-up period will end if you enroll on another protocol or start receiving standard therapy.

# **CONFLICT OF INTEREST (COI)**

The NIH reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

No NIH investigator involved in this study receives payments or other benefits from any company whose drug, product or device is being tested.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor, NCI Cancer Therapy Evaluation Program (CTEP), or their agent(s)
- Designated investigators from other cancer centers participating in this study, including the University of Southern California/Norris Comprehensive Cancer Center; the University of California, Davis, Cancer Center; and Stanford University Medical Center.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

# POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Alice P. Chen, chenali@mail.nih.gov, 240-781-3320. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

# **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


IRB NUMBER: 13C0044 IRB APPROVAL DATE: 04/06/2021

| - | I have read the explanation about this study arns. I consent to participate in this study. | 0 11 |
|---|---|---|
| Signature of Research Particip | ant Print Name of Research P | articipant Date |
| about this study and have been<br>to make research decisions on | ntative (LAR) for an Adult Unable to Corn given the opportunity to discuss it and to ask behalf of the adult participant unable to consercable, the information in the above consent was to participate in the study. | questions. I am legally authorized and have the authority to provide |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | r Date |
| Signature of Witness* | Print Name of Witness | Date |
| INTERPRETER: An interpreter, or other in | SECTION TO BE COMPLETED REC<br>dividual, who speaks English and the participal<br>dividual, and served as a witness. The invest | ant's preferred language facilitat |
| An interpreter or other in | dividual, who speaks English and the participal consent but <u>did not</u> serve as a witness. The n | |
| | is: | · |


CC pre rCR ICF template v. 05.05.2020